CLINICAL TRIAL: NCT05944081
Title: Multicenter, Not Randomised, Non-interventional, Postmarket Clinical Follow-Up (PMCF) Study on the Performance / Safety of Arcadius XP L® Interbody Fusion Device
Brief Title: Postmarket Clinical Follow-Up Study on Arcadius XP L® Interbody Fusion Device
Acronym: ARREST
Status: Withdrawn | Type: Observational
Why Stopped: Limited patient willingness and clinic capacity hindered follow-up data collection for the registry study, as appointments required extra resources beyond routine care.
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2110
Record Dates: First submitted 2023-07-03; First posted 2023-07-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low-back Pain; Degenerative Disc Disease; Spondylolysis Lumbar; Postdiscectomy Syndrome; Posttraumatic Instability
Keywords: stand-alone cage; lumbar spine; interbody fusion device
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arcadius XP L®: all patients who received a Arcadius XP L® interbody fusion device between 2016 until approx. January 2021 (minimum Follow-up is one year) in the study center
  Interventions: Device: ArcadiusXP L® Interbody Fusion System

INTERVENTIONS:
Device: ArcadiusXP L® Interbody Fusion System — The ArcadiusXP L® Interbody Fusion System is a stand-alone device intended to be used with four bone screws if no supplement fixation is used to stabilize the lumbar spine through an anterior approach. Levels of anterior lumbar interbody fusion for the indications listed in the instructions for use are from L2-S1.

SUMMARY:
The purpose of this study is to collect clinical and radiological mid-term (min. 1 year) data on the ArcadiusXP L® lumbar stand-alone cage in a post-market clinical follow-up study (PMCF) limited to 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients who received a Arcadius XP L® interbody fusion device between 2016 until approx. January 2021 (minimum Follow-up is one year) in the study center
* all indications as given by the instructions for use: degenerative disc disease (DDD), Instability, Spondylolisthesis up to grade 1, Post-discectomy syndrome, Post-traumatic instability
* Written informed consent for the documentation of clinical and radiological results

Exclusion Criteria:

* Patient is not willing or able to participate at the follow-up examination
* Patients living outside a radius of 100 km around the study center
* all contraindications as given by the instructions for use:

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients that received an Arcadius XP L® interbody fusion device in accordance with the indications given in the instructions for use:
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome after minimum 1 year postoperatively | at follow-up approximately 1 year postoperatively
  The Oswestry Disability Index (ODI) is designed to measure back-specific disability. The questionnaire is self-administered and has 10 items concerning pain and activities of daily living including personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. It is a self-administered questionnaire Each section is scored on a 0-5 scale, 5 is for maximum disability. The index is calculated by dividing the total score by the total possible score, which is multiplied by 100 and expressed as a percentage. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Pain assessment | at follow-up approximately 1 year postoperatively
  Pain will be assessed by the patient using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal/worst pain". Pain will be recorded at minimum 12 months postoperatively, if available in the preoperative clinical routine data, it will also be recorded in the study.
Development Quality of life (EQ-5D-5L) | at follow-up approximately 1 year postoperatively
  "EQ-5D-5L" is a standardized 5-dimension 5-level measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. In order to analyze the quality of life of the patients, the EQ-5D-5L is used. The score is self-completed by the patient and will therefore be used in German.
Radiological Outcome: Bone fusion | at follow-up approximately 1 year postoperatively
  After Interbody Fusion surgery fusion of the treated segment is aspired. Thus, the implant design shall allow on-/ingrowth to/into the material. The fusion status can be determined from radiographs (static or dynamic). Bony fusion can be characterized quantitatively by the fusion rate.
Rate of (Serious) adverse events | at follow-up approximately 1 year postoperatively
  Occurrence of complications potentially associated with the implanted devices can never be fully excluded during spinal surgery. In order to monitor potential complication and to identify so far unknown complications AEs and SAEs deemed related to the investigational device are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Reithmeier, Dr., Principal Investigator — Schelztor-Klinik
Locations (3):
- Germany (3):
  - Schelztor-Klinik Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Medius Klinik Nürtingen, Nürtingen, Baden-Wurttemberg
  - Rems-Murr-Klinik Schorndorf, Schorndorf, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: No